CLINICAL TRIAL: NCT03016468
Title: A Multicenter, 16-Week, Open-label Study Evaluating the Safety of Transition From Selexipag to Remodulin® Then Oral Treprostinil in Symptomatic Subjects With Pulmonary Arterial Hypertension
Brief Title: Safety of Transition From Selexipag to Remodulin® Then Oral Treprostinil in Symptomatic Adult PAH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-207
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Oral Treprostinil; Remodulin; Selexipag; 6 Minute Walk Test
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Parenteral Remodulin then Oral Treprostinil (Experimental)
  Interventions: Drug: Parenteral Remodulin (treprostinil) injection; Drug: Oral Treprostinil

INTERVENTIONS:
Drug: Parenteral Remodulin (treprostinil) injection — Remodulin will be provided in vial strengths of 1, 2.5, 5, and 10 mg/mL. Subjects will be admitted to the hospital and IV Remodulin will be initiated within 12 hours after the last dose of selexipag. Subjects will remain under observation in the inpatient setting for at least the first 72 hours of Remodulin administration. Subjects will be transitioned to an equivalent dose of SC Remodulin at discharge.
  Other Names: Remodulin
Drug: Oral Treprostinil — Oral treprostinil will be provided as 0.125-, 0.25-, 1-, or 2.5-mg extended-release tablets. Oral treprostinil will be dosed three times daily with food.
  Other Names: Orenitram

SUMMARY:
This is a multicenter, single-arm trial to evaluate the safety of the transition from Selexipag to Remodulin® then Oral Treprostinil in Symptomatic Subjects with Pulmonary Arterial Hypertension (PAH). The study will include about 30 subjects at approximately 10 clinical trial centers. The treatment phase of the study will last approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of symptomatic idiopathic or heritable PAH, PAH associated with connective tissue disease, PAH associated with HIV infection, PAH associated with repaired congenital systemic-to-pulmonary shunt (at least 1 year since repair with respect to the date of providing informed consent), or PAH associated with appetite suppressant or toxin use.
2. The subject must be classified as WHO FC II or III at Baseline.
3. The subject is receiving selexipag for the treatment of WHO Group 1 PAH for a minimum of 90 days from Baseline.
4. Subject is in need of escalation of therapy, as determined by the Investigator.
5. Subject must be receiving a Food and Drug Administration (FDA)-approved PDE5-I or sGC stimulator and/or an ERA and has been at the current stable dose for at least 28 days prior to Baseline.

Exclusion Criteria:

1. The subject is receiving selexipag for any other disease or condition other than the treatment of WHO Group 1 PAH.
2. The subject has a Baseline 6MWD of less than 150 meters.
3. The subject's Baseline 6MWD has decreased more than 40% from the pre-selexipag baseline.
4. The subject has a history of ischemic heart disease (defined as either symptomatic or requiring anti-anginal therapy or experienced a documented myocardial infarction within the previous 6 months of Baseline), or a history of left sided myocardial dysfunction as evidenced by a PAWP greater than 15 mmHg or a left ventricular ejection fraction less than 40%.
5. The subject has previously been treated with any parenteral prostacyclin or oral treprostinil for a period of 90 days or more.
6. The subject has a history of 1 or more of the following signs of relevant lung disease within 180 days before Baseline:

   1. Total lung capacity less than 60% of predicted normal.
   2. Forced expiratory volume in 1 second is less than 55% of predicted normal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) through 16 Weeks | 16 Weeks

SECONDARY OUTCOMES:
Change in 6-minute Walk Distance (6MWD) from Baseline to Week 16 | Baseline and Week 16
Change in Borg Dyspnea Score Immediately After 6-minute Walk Test (6MWT) from Baseline to Week 16 | Baseline and Week 16
Change in plasma concentration of N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) from Baseline to Week 16 | Baseline and Week 16
Change in Pulmonary Arterial Hypertension (PAH) Symptoms Score from Baseline to Week 16 | Baseline and Week 16
Change in Score on Treatment Satisfaction Questionnaire for Medication (TSQM) from Baseline to Week 16 | Baseline and Week 16